CLINICAL TRIAL: NCT04934189
Title: Empowerment Self-Defense Training for the Prevention of Victimization of Transgender Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Danielle Berke, Assistant Professor, Hunter College of City University of New York
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: R21MD014807 (NIH); 5R21MD014807-02 (NIH)
Record Dates: First submitted 2021-06-04; First posted 2021-06-22 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Violence, Sexual
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: The proposed curriculum will be systematically refined based on delivery of the intervention to 3 groups of 16 TW each in a 20-hour training program, in 5 4-hour sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial (Other): Refinement and assessment of the feasibility and acceptability of the Empowerment Self-Defense curriculum will occur in Phase 2 through the delivery of the tailored ESD curriculum to 3 groups of 16 TW.
  Interventions: Behavioral: Empowerment Self Defense Training

INTERVENTIONS:
Behavioral: Empowerment Self Defense Training — We have contracted with Prepare, Inc., the New York City chapter of IMPACT International to deliver the tailored ESD violence prevention intervention. IMPACT is an international ESD violence prevention organization with chapters across the United States. Prepare, Inc. will provide facilitators who have completed IMPACT's nationally standardized ESD violence prevention program requirements that include receipt of over 100 hours of training. IMPACT training is open to trans and cisgender women. The extensive training of IMPACT facilitators promotes intervention efficacy, while the risk of potential bias conferred by their experience with a pre-existing curriculum is mitigated by our community-engaged approach (i.e.,TW community members, service providers, and scientists [PI and Co-I] collectively shape the content of the final tailored ESD intervention, and TW co-facilitators will be present in every training session).

SUMMARY:
The proposed project aims to develop and refine a tailored Empowerment Self Defense (ESD) violence prevention training for diverse TW through a series of sequential Aims: a) develop an initial draft of an ESD violence prevention curriculum tailored to TW (Aim 1); b) evaluate the feasibility and acceptability of recruitment, assessment procedures, retention and follow-up procedures, and implementation of the new intervention (Aim 2); and c) assess the preliminary efficacy of the tailored intervention program to increase use of self-protective resistance strategies, mitigate minority stressors and attitudinal barriers to self-defense, and reduce rates of exposure to violence (Exploratory Aim).

The investigators will accomplish these aims using a two-phase research design that begins with formative qualitative work engaging research partners on a community board and a small sample of research participants. Information for Phase 1 can be located in Protocol number 2020-0017. Further refinement and assessment of the feasibility and acceptability of the curriculum using Phase 1 findings will occur in Phase 2 through the delivery of the tailored ESD curriculum to 3 groups of 16 TW. To assess the preliminary efficacy of the tailored intervention, program participants will complete a battery of validated questionnaires assessing use of resistance strategies, gender-minority and general psychological factors hypothesized to mediate the behavioral effects of the intervention, and exposure to victimization experiences prior to, immediately following, and 6 months post-completion of the training. Together, the proposed research will lay the foundation for a large-scale randomized controlled trial (RCT) of the tailored ESD violence prevention curriculum.

DETAILED DESCRIPTION:
This study leverages the strong evidence-base for Empowerment Self-Defense (ESD) violence prevention to address disparities in violence exposure among TW. The overarching goal of this R21 is to develop and refine a tailored ESD violence prevention training for diverse TW through a series of sequential Aims: a) develop an initial draft of an ESD violence prevention curriculum tailored to TW (Aim 1); b) evaluate the feasibility and acceptability of recruitment, assessment procedures, retention and follow-up procedures, and implementation of the new intervention (Aim 2); and c) assess the preliminary efficacy of the tailored intervention program to increase use of self-protective resistance strategies, mitigate minority stressors and attitudinal barriers to self-defense, and reduce rates of exposure to violence (Exploratory Aim). Together, the proposed research will lay the foundation for a large-scale randomized controlled trial (RCT) of the tailored ESD violence prevention curriculum. The investigators will accomplish these aims using a two-phase research design that begins with formative qualitative work engaging research partners on a community board and a small sample of research participants. This data will be used to inform the development and refinement of the ESD violence prevention curriculum for TW. Further refinement and assessment of the feasibility and acceptability of the curriculum will occur in Phase 2 through the delivery of the tailored ESD curriculum to 3 groups of 16 TW. To assess the preliminary efficacy of the tailored intervention, program participants will complete a brief survey assessing the program directly after completion, as well as a battery of validated questionnaires assessing use of resistance strategies, gender-minority and general psychological factors hypothesized to mediate the behavioral effects of the intervention, and exposure to victimization experiences prior to, immediately following, and 6 months post-completion of the training.

The overall goal of this study is to use findings from Phase 1 to deliver and refine a tailored ESD violence prevention training for diverse trans women.

Participants for Phase 2 (n = 48) will be recruited from online forums including social media sites (e.g., Facebook, Twitter), banner ads on social networking/dating sites (e.g., Scruff, BGC Live, OK Cupid, Lex) that are trans-inclusive and through dissemination of paper and/or electronic recruitment flyers with leaders of community organizations that connect transgender individuals (e.g., AVP; Callen Lorde, Trans-lantinx network). Participants from prior studies who consented to future contact will be sent the study flyer by email.

The proposed curriculum will be systematically refined based on delivery of the intervention to 3 groups of 16 TW each in a 20-hour training program, in 5 4-hour sessions. The investigators have contracted with Prepare, Inc., the New York City chapter of IMPACT International to deliver the tailored ESD violence prevention intervention. IMPACT is an international ESD violence prevention organization with chapters across the United States. Prepare, Inc. will provide facilitators who have completed IMPACT's nationally standardized ESD violence prevention program requirements that include receipt of over 100 hours of training. IMPACT training is open to trans and cisgender women. The extensive training of IMPACT facilitators promotes intervention efficacy, while the risk of potential bias conferred by their experience with a pre-existing curriculum is mitigated by our community-engaged approach (i.e.,TW community members, service providers, and scientists [PI and Co-I] collectively shape the content of the final tailored ESD intervention, and TW co-facilitators will be present in every training session). Prior to the start of group, facilitators will review the tailored curriculum in detail and attend 2-3 supervision/training meetings with the PI. These meetings will consist of reviewing the curriculum, role-plays of critical intervention components, and discussion of questions or concerns.

The primary outcome of Aim 2 is to evaluate our ability to recruit our target (n = 48) and retain >75% over the course of the intervention. Successful completion of the pilot trial, including meeting or exceeding these benchmarks for success, will determine the feasibility and acceptability of recruiting participants into a future RCT. Preliminary efficacy of the tailored ESD violence prevention intervention will be evaluated as an exploratory aim. Participants enrolled in the pilot trial will be administered a battery of validated baseline questionnaires at baseline, immediately following the course, and 6 months after course completion including:

* Demographics
* Social Class Ladder
* Community Ladder
* Service Utilization Form
* Sexual experiences Survey
* Everyday Discrimination Scale
* Conflict Tactics Scale
* Gender Minority Stress Risk and Resilience Scale
* Post Traumatic Stress Disorder Symptom Checklist for DSM-5 (PCL-5)
* Sexual Assertiveness Questionnaire
* Resistance Tactics Survey
* Dating Self-Protection
* Illinois Rape Myth Acceptance
* Resistance Self-Efficacy
* Personal Progress
* Transgender Congruence Scale
* Depression Anxiety and Stress Scale
* Quick Drinking Screen
* DAST-10

Brief acceptability checklists will be administered after each course session, which will contain a brief list of topics covered during that training session and participants will indicate which of the topics participants felt were adequately covered. Lastly, an exit interview will be scheduled on the final day of the course, and will take place over the weeks immediately following the completion of the course. Interviews will be video recorded using the Zoom videoconferencing platform. The video-recorded qualitative interviews will be recorded and transcribed verbatim using the Zoom transcription function (omitting identifying information) and verified for accuracy.

The investigators will use three strategies to improve retention, based on an intensive evidence-based follow-up protocol with which the PI has considerable experience. First, participants will be compensated for completion of the assessment appointments at increasing increments over time. Second, at baseline, participants will be asked to provide extensive locating information and to provide names of two local persons to be contacted in the event that the participant cannot be reached. This information will be updated at the time of follow-up survey administration. Third, participants will receive cash for each of the five session acceptability checklists the participants complete.

Analyses will be of two primary types: (a) examinations of whether feasibility targets were met across a variety of measures; and (b) examinations of the efficacy of the tailored ESD violence prevention intervention. The investigators will use repeated measures one-way ANOVA to test if the tailored ESD curriculum has statistically significant effect on measures of behavioral and psychological/attitudinal change. If a significant effect is detected, the investigators will use Tukey's pairwise-comparison procedure to compare all treatment means, with a 95% family confidence coefficient. To assess changes in exposure to victimization, the investigators will collapse into three levels: (a) no history of victimization; (b) moderate victimization; (c) severe victimization. For this categorical data, a chi-square test of independence will be performed to compare posttreatment vs. pre-treatment, and 6-month FU vs. pre-treatment respectively to assess the preliminary efficacy of the program, with a family-wise type I error controlled at 0.05 using Bonferroni procedure. Our efficacy outcomes are exploratory and powered to detect large effect sizes. In the largest scale RCT of an ESD violence prevention program to date, rates of completed assault among women receiving resistance training were reduced by half at 1-year follow-up. However, as there are no existing studies that report on ESD efficacy among TW, the investigators will use results of our exploratory efficacy analysis to shape power analyses for a subsequent, fully powered, RCT.

ELIGIBILITY:
Inclusion Criteria:

* Transgender women (i.e., male assigned at birth, currently identified on the transfeminine spectrum)
* Between the ages of 18 and 65.

Exclusion Criteria:

* Cisgender men and women
* Transgender men

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women (i.e., male assigned at birth, currently identified on the transfeminine spectrum) between the ages of 18 and 65. This inclusion criteria is necessary to iteratively tailor and finalize the adapted ESD violence prevention program for transgender women.
Enrollment: 62 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle S Berke, Principal Investigator — Hunter College of The City University of New York
Locations (1):
- Hunter College, City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith AM, Hotchkiss M, Gilbert C, Williams DN, Madhav K, Bloomfield K, Pautz CR, Berke DS. Process adaptations to community-engaged research for preventing victimization against trans women: Failure as a blueprint toward nonexploitative implementation science. Am Psychol. 2023 Feb-Mar;78(2):186-198. doi: 10.1037/amp0001063. PMID 37011169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were adults recruited from the community between July 2021 and November 2021. Participants were recruited through advertisements on social media and via email flyers distributed to community organizations and leaders. Recruitment materials (advertisements and flyers) advertised a no cost group Empowerment Self-Defense program for Trans Women and Trans Femmes and indicated that participants would be compensated up to $230.
Pre-assignment Details: Participants were excluded from analyses if they did not meet inclusion/exclusion criteria; met screening criteria but did not respond to enrollment invitation; replied to enrollment invitation emails but did not complete baseline survey and never attended class; completed baseline survey but missed the first three consecutive sessions (i.e., dropped out). Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Period: Overall Study
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Started | 60
Completed | 39
Not Completed | 21
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 17

BASELINE CHARACTERISTICS:
Population: We contracted with Prepare, Inc. to provide the ESD group intervention. Prepare facilitators recommended a maximum of 16 participants per group to ensure the provision of adequate space and attention to each participant. Thus 3 groups were needed to simultaneously achieve target recruitment and provision of an "adequate treatment dose" to all participants. As all participants received the same treatment dose, results were analyzed in a single treatment arm pre-post design.
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.59 (12.76)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transwomen/Trans femmes | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 17
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 39
Annual Household Income [Count of Participants; unit: Participants]
  under $10,000 | 21
  $10,001-$20,000 | 8
  $20,001- $30,000 | 4
  $40,0001-$50,000 | 3
  $70,001-$80,000 | 1
  $90,000-$100,000 | 1
  over $150,000 | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Rating on Sexual Assertiveness at Baseline
Description: The Sexual Assertiveness Questionnaire uses a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Higher scores are indicative of more impaired assertiveness. The measure comprises a 14-item Relational Sexual Assertiveness subscale and consists of items such as "I worry that my partner won't like me unless I engage in sexual behavior" and "I am easily persuaded to engage in sexual activity" and a 7-item Confidence and Communication subscale. A sample item is "I lack confidence in sexual situations." A total score was created by taking the average of all 14 items (range = 1-5).
Time Frame: Baseline
Population: Syntax was generated in SPSS to calculate the baseline mean response across the 14-item measure for all respondents providing data for at least two of the scale items. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale | 2.77 (1.15)

2. Primary Outcome: Change in Sexual Assertiveness From Baseline to 3 Month Followup
Description: as for outcome 1
Time Frame: Change from Baseline at 3 months
Population: Syntax was generated in SPSS to calculate the posttreatment mean response across the 14-item measure for all respondents providing data for at least two of the scale items. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale | 2.47 (1.18)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 3-month) mean was statistically different from the baseline mean; Test type: Other; p = .08, t-test, 1 sided; Mean Difference (Final Values) = .295, Standard Deviation 1.184

3. Primary Outcome: Change in Sexual Assertiveness From Baseline to 6 Month Follow up
Description: as for outcome 1
Time Frame: Change from Baseline at 6 months
Population: Syntax was generated in SPSS to calculate the mean response across the 14-item measure for all respondents providing data for at least two of the scale items during the 6 month follow-up assessment period. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale | 2.44 (0.86)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month follow-up mean) was statistically different from the baseline mean; Test type: Other; p = .005, t-test, 1 sided; Mean Difference (Net) = .417, Standard Deviation .89

4. Primary Outcome: Average Number of Resistance Tactics Endorsed at Baseline
Description: The Resistance Tactics Questionnaire will be used to measure participants use of six self-defense strategies via "yes" or "no" responses to the question prompt. The self-defense strategies assessed included (a) assertive body language (e.g., walking confidently), (b) assertive verbal responses (e.g., saying "no"), (c) avoiding telegraphing emotions (e.g., providing an assertive verbal response even when nervous), (d) attention to your intuition (e.g., trusting your gut), (e) yelling and running, and (f) physical self-defense. Higher scores indicate greater use of resistance tactics. A total score was created by calculating the sum of all 6 items (range: 0-6).
Time Frame: Baseline
Population: Syntax was generated in SPSS to calculate the baseline mean response across the 6-item measure for all respondents providing data for at least two of the scale items. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 4.31 (1.76)

5. Primary Outcome: Change in Resistance Tactics From Baseline to 3 Month Follow up
Description: as for outcome 4
Time Frame: Change from Baseline at 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 4.41 (1.87)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.40, t-test, 1 sided; Mean Difference (Net) = -.103, Standard Deviation 2.500

6. Primary Outcome: Change in Resistance Tactics From Baseline to 6 Month Follow up
Description: as for outcome 4
Time Frame: Change from Baseline and 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 33
score on a scale | 4.34 (1.78)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month follow-up) mean was statistically different from the baseline mean; Test type: Other; p = .49, t-test, 1 sided; Mean Difference (Net) = -.01, Standard Deviation 2.08

7. Primary Outcome: Average Use of Dating Self-Protection Against Rape Strategies at Baseline
Description: Participant's use of protective strategies against sexual victimization will be assessed with the Dating Self-Protection Against Rape Scale. Participants will report the frequency with which they engage in a series of 15 behaviors used to for self-protection (e.g., "How often do you pay attention to your dating partner's drug/alcohol intake?"). Responses are provided along a 6-point scale ranging from never to always. Higher scores indicate greater use of self-protective strategies. A total score was created by calculating the average of all 15 items (range: 1-6).
Time Frame: Baseline
Population: Syntax was generated in SPSS to calculate the baseline mean response across the 15-item measure for all respondents providing data for at least two of the scale items. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 35
score on a scale | 3.64 (1.12)

8. Primary Outcome: Change in Dating Self-Protection Against Rape From Baseline to 3 Month Follow up
Description: Participant's use of protective strategies against sexual victimization will be assessed with this scale. Participants will report the frequency with which they engage in a series of 15 behaviors used to for self-protection (e.g., "How often do you pay attention to your dating partner's drug alcohol intake?"). Responses are provided along a 6-point scale ranging from never to always. Higher scores indicate greater use of self-protective strategies. A total score was created by calculating the average of all 15 items (range: 1-6).
Time Frame: Change from Baseline at 3 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 35
score on a scale | 3.44 (1.26)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .21, t-test, 1 sided; Mean Difference (Net) = .195, Standard Deviation 1.41

9. Primary Outcome: Change in Dating Self-Protection Against Rape From Baseline to 6 Month Follow up
Description: Participant's use of protective strategies against sexual victimization will be assessed with the Dating Self-Protection Against Rape Scale. Participants will report the frequency with which they engage in a series of 15 behaviors used to for self-protection (e.g., "How often do you pay attention to your dating partner's drug alcohol intake?"). Responses are provided along a 6-point scale ranging from never to always. Higher scores indicate greater use of self-protective strategies. A total score was created by calculating the average of all 15 items (range: 1-6).
Time Frame: Change from Baseline at 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale | 3.68 (1.19)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean was statistically different from the baseline mean; Test type: Other; p = .47, t-test, 1 sided; Mean Difference (Net) = .019, Standard Deviation 1.43

10. Secondary Outcome: Average Endorsement of Rape Myth Acceptance at Baseline Scale
Description: The 45-item scale Illinois Rape Myth Acceptance Scale assesses the endorsement of rape myth attitudes supportive of sexual coercion and aggression. Rape myths include "beliefs about rape (i.e., about its causes, context, consequences, perpetrators, victims, and their interaction) that serve to downplay, or justify sexual violence that men commit again women" (Gerger et al., 2007). The scale is formatted on a 7-point Likert-type scale ranging from "1" (strongly disagree) to "7" (strongly agree). A total score was created by calculating the average rating across all 45-items (range: 1-7).
Time Frame: Baseline
Population: Syntax was generated in SPSS to calculate the baseline mean response across the 45-item measure for all respondents providing data for at least two of the scale items. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 1.81 (.915)

11. Secondary Outcome: Change in Rape Myth Acceptance From Baseline to 3 Month Follow up
Description: The Illinois Rape Myth Acceptance Scale is a 45-item scale assessing the endorsement of rape myth attitudes supportive of sexual coercion and aggression. Rape myths include "beliefs about rape (i.e., about its causes, context, consequences, perpetrators, victims, and their interaction) that serve to downplay, or justify sexual violence that men commit against women" (Gerger et al., 2007). The scale is formatted on a 7-point Likert-type scale ranging from "1" (strongly disagree) to "7" (strongly agree). A total score was created by calculating the average rating across all 45-items (range: 1-7). Higher scores indicate greater endorsement of rape myths.
Time Frame: Change from Baseline at 3 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 1.64 (.827)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .16, t-test, 1 sided; Mean Difference (Net) = .175, Standard Deviation 1.02

12. Secondary Outcome: Change in Rape Myth Acceptance From Baseline to 6 Month Follow up Scale
Description: This 45-item Illinois Rape Myth Acceptance Scale assesses the endorsement of rape myth attitudes supportive of sexual coercion and aggression. Rape myths include "beliefs about rape (i.e., about its causes, context, consequences, perpetrators, victims, and their interaction) that serve to downplay, or justify sexual violence that men commit against women" (Gerger et al., 2007). The scale is formatted on a 7-point Likert-type scale ranging from "1" (strongly disagree) to "7" (strongly agree). Higher scores indicate greater endorsement of rape myths. A total score was created by calculating the average rating across all 45-items (range: 1-7).
Time Frame: Change from Baseline at 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale | 1.78 (.794)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = .38, t-test, 1 sided; Mean Difference (Net) = .0481, Standard Deviation .926

13. Secondary Outcome: Baseline Average Rating of Resistance Self-Efficacy
Description: Participants' confidence in utilizing assertive responses to potentially threatening dating situations was assessed by seven items on the Resistance Self-Efficacy Scale (i.e., "If someone you were with was attempting to get you to have sex with them and you were not interested, how confident are you that you could successfully resist their advances?"; Marx, Calhoun, Wilson, & Meyerson, 2001; Ozer & Bandura, 1990). Responses are provided along a 7-point scale, ranging from not at all confident to very confident. Higher scores indicate great resistance self-efficacy. A total score was created by calculating the average rating across all items (range: 1-7).
Time Frame: Baseline
Population: Syntax was generated in SPSS to calculate the baseline mean response across the 7-item measure for all respondents providing data for at least two of the scale items. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 4.59 (1.64)

14. Secondary Outcome: Change in Resistance Self-Efficacy From Baseline to 3 Month Follow up
Description: as for outcome 13
Time Frame: Change from Baseline at 3 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 4.41 (1.93)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .35, t-test, 1 sided; Mean Difference (Net) = .179, Standard Deviation 2.73

15. Secondary Outcome: Change in Resistance Self-Efficacy From Baseline to 6 Month Follow up
Description: Participants' confidence in utilizing assertive responses to potentially threatening dating situations was assessed by seven items on the Self-Efficacy Scale (i.e., "If someone you were with was attempting to get you to have sex with them and you were not interested, how confident are you that you could successfully resist their advances?"; Marx, Calhoun, Wilson, & Meyerson, 2001; Ozer & Bandura, 1990). Responses are provided along a 7-point scale, ranging from not at all confident to very confident. Higher scores indicate great resistance self-efficacy. A total score was created by calculating the average rating across all items (range: 1-7).
Time Frame: Change from Baseline at 6 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale | 5.04 (1.65)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = .17, t-test, 1 sided; Mean Difference (Net) = -.335, Standard Deviation 2.05

16. Secondary Outcome: Average Rape Attribution at Baseline
Description: Participants attributions of blame following experiences of sexual victimization will be assessed by 25 items on the Rape Attribution Scale (Frazier, 2002; Frazier & Seales, 1997). Responses are provided along a 5-point scale, ranging from never to very often, whereby higher scores indicate higher levels of blame. Five subscales will be utilized to explore various attributions of blame, including (a) societal blame, (b) behavioral selfblame, (c) characterological self-blame, (d) chance, and (e) rapist blame. A total score was to be created by calculating the average rating across all items (range: 1-5).
Time Frame: Baseline
Population: data not collected since this measure was inadvertently omitted from the baseline and follow-up measurement battery administered to participants enrolled in the clinical trial
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 0

17. Secondary Outcome: Change in Rape Attribution From Baseline to Follow up Assessments
Description: as for outcome 16
Time Frame: Change from 3 months at 6 months
Population: as for outcome 16
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 0

18. Secondary Outcome: Average Rating of Gender Identity Non-Affirmation, Internalized Transphobia, Concealment, Community Connectedness, and Pride
Description: Designed for use with transgender and gender nonconforming people, the Gender Minority Stress and Resilience measure is one of the few that assesses gender identity-related constructs. It was designed to take into account unique gender minority distal stressors as was a resilience factors. These subscales will be used in this current study to test hypothesized mediators of the effects of the ESD violence prevention training on behavioral outcomes. Responses are given on a a 5-point Likert response scale (Strongly Disagree to Strongly Agree). Higher scores are indicative of greater phenomena. Six subscale scores were created by calculating the average rating for measure items corresponding with each construct: nonaffirmation of transgender identity, internalized transphobia, identity nondisclosure, negative expectations, community connection, and pride. Range for all subscales: 1-5
Time Frame: Baseline
Population: Syntax was generated in SPSS to calculate the baseline mean response across each subscale measuring nonaffirmation of transgender identity, internalized transphobia, identity nondisclosure, negative expectations, community connection, and pride respectively for all respondents providing data for at least two of the scale items on each subscale. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale
  Nonaffirmation | 1.78 (1.06)
  Internalized Transphobia | 0.96 (.86)
  Identity Nondisclosure | 1.76 (1.37)
  Negative Expectations | 1.88 (1.35)
  Community Connection | 2.12 (1.18)
  Pride | 2.03 (1.12)

19. Secondary Outcome: Change in Non-Affirmation, Internalized Transphobia, Concealment, Community Connectedness, and Pride From Baseline to 3 Month Follow up
Description: as for outcome 18
Time Frame: Change from Baseline at 3 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale
  Nonaffirmation | 1.41 (0.89)
  Internalized Transphobia | 0.77 (0.79)
  Identity Nondisclosure | 1.72 (1.40)
  Negative Expectations | 2.05 (1.35)
  Community Connection | 2.20 (0.83)
  Pride | 1.75 (1.38)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 3-month followup) mean for gender nonaffirmation was statistically different from the baseline mean; p = .02, t-test, 1 sided — A priori threshold for statistical significance was <.05; t-test = 2.18
Statistical Analysis 2: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 3-month followup) mean for internalized transphobia was statistically different from the baseline mean; p = .10, t-test, 1 sided — A priori threshold for statistical significant was p <.05; t-test = 1.29
Statistical Analysis 3: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 3-month followup) mean for identity nondisclosure was statistically different from the baseline mean; p = .43, t-test, 1 sided — A priori threshold for statistical significance was p < .05; t-test = 0.17
Statistical Analysis 4: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 3-month followup) mean for negative expectations was statistically different from the baseline mean; p = .25, t-test, 1 sided — A priori threshold for statistical significance was p < .05; t-test = -.68
Statistical Analysis 5: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 3-month followup) mean for community connection was statistically different from the baseline mean; p = .36, t-test, 1 sided — The a priori threshold for statistical significance was p < .05; t-test = -.36
Statistical Analysis 6: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 3-month followup) mean for pride was statistically different from the baseline mean; p = .47, t-test, 1 sided — The a priori threshold for statistical significance was p < .05; t-test = -.09

20. Secondary Outcome: Change in Gender Identity Non-Affirmation, Internalized Transphobia, Concealment, Community Connectedness, and Pride From Baseline to 6 Month Follow up
Description: as for outcome 18
Time Frame: Change from Baseline at 6 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 34
score on a scale
  Nonaffirmation | 1.28 (0.96)
  Internalized Transphobia | 0.69 (0.63)
  Identity Nondisclosure | 1.57 (1.02)
  Negative Expectations | 1.69 (1.08)
  Community Connection | 2.20 (0.95)
  Pride | 2.00 (1.11)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean for gender nonaffirmation was statistically different from the baseline mean; p < .001, t-test, 1 sided — The a priori threshold for statistical significance was p < .05; t-test = 3.76; A series of one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean was statistically different from the baseline mean for each of the five gender minority stress subscales measured. See below for T-scores and associated p-values for each statistical test. Nonaffirmation (t = 3.76; p = .001) Internalized Transphobia (t = 2.01; p = .02) Negative Expectations (t = 2.06; p =.02) Community Connection (t = -0.82; p =.21) Pride (t = .01; p = .50 )
Statistical Analysis 2: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean for internalized transphobia was statistically different from the baseline mean; p = .02, t-test, 1 sided — The a priori threshold for statistical significance is p < .05; t-test = 2.01
Statistical Analysis 3: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean for identity nondisclosure was statistically different from the baseline mean; p = .06, t-test, 1 sided — The a priori threshold for statistical significance was p < .05; t-test = 1.61
Statistical Analysis 4: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean for negative expectations was statistically different from the baseline mean; p = .02, t-test, 1 sided — The a priori threshold for statistical significance was p < .05; t-test = 2.06
Statistical Analysis 5: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean for community connection was statistically different from the baseline mean; p = .21, t-test, 1 sided — The a priori threshold for statistical significance was p < .05; t-test = -.818
Statistical Analysis 6: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month followup) mean for pride was statistically different from the baseline mean; p = .50, t-test, 1 sided — The a priori threshold for statistical significance was p < .05; t-test = .009

21. Secondary Outcome: Percentage of Participants Endorsing Rape, Sexual Assault, and No Sexual Victimization at Baseline
Description: The Sexual Experience Survey Short Form Victimization (SES-SFV) is the most widely used measure in sexual assault research. A primary strength of the measure is that it does not require participant to label their experiences as "sexual assault" or "rape." Rather, it utilizes a series of 10 sexually explicit questions that assess t past sexual behavior along a variety of dimensions. Experiences can be classified as "completed rape," "attempted rape," "coercion," "attempted coercion," or "nonconsensual sexual contact." Participants were assigned a score of "0" if they denied the question and a score of "1" if they endorsed the question. Participants with a score of 0 for all items were categorized as having no history of victimization. Participants with a score of 1 for any item assessing sexual coercion or nonconsensual sexual contact were categorized as having experienced sexual assault. Participants with a 1 for any rape item were catagorized as having experienced rape.
Time Frame: Baseline
Population: To assess rates of exposure to sexual victimization we collapsed participants response into three dichotomous variable levels: 1) no history of victimization; 2) history of moderate victimization (non-penetrative assault); and 3) history of severe victimization (penetrative assault). Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 37
Participants
  Rape | 9
  Sexual Assault | 9
  No Victimization | 19

22. Secondary Outcome: Change in Percentage of Participants Endorsing Rape, Sexual Assault, and No Victimization From Baseline to 3 Month Followup
Description: as for outcome 21
Time Frame: Change from Baseline at 3 months
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
Participants
  Rape | 7
  Sexual Assault | 7
  No Victimization | 22

23. Secondary Outcome: Change in Percentage of Participants Endorsing Rape, Sexual Assault, and No Victimization From Baseline to 6 Month Followup
Description: as for outcome 21
Time Frame: Change from Baseline at 6 months
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
Participants
  Rape | 5
  Sexual Assault | 7
  No Victimization | 24
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; For this categorical data, chi-square tests of independence were performed to compare post-treatment (i.e., 3 month followup) vs 6 month followup numbers of participants reporting freedom from sexual victimization over a 6 month time period; Test type: Other; p = .04, Chi-squared — A priori threshold for statistical significance was p <.05; Chi-squared = 5.59
Statistical Analysis 2: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — For this categorical data, chi-square tests of independence were performed to compare post-treatment (i.e., 3 month followup) vs 6 month followup numbers of participants reporting any exposure to nonpenetrative sexual assault over a 6 month time period; p = .55, Chi-squared — A priori threshold for statistical significance was p < .05; Chi-squared = .21
Statistical Analysis 3: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; Test type: Other — For this categorical data, chi-square tests of independence were performed to compare post-treatment (i.e., 3 month followup) vs 6 month followup numbers of participants reporting exposure to rape over a 6 month time period; p = .59, Chi-squared — A priori threshold for statistical significance was p < .05; Chi-squared = .11

24. Secondary Outcome: Baseline Average Likelihood of Endorsing Gender-Based Victimization
Description: This subscale of the Gender Minority Stress and Resilience Measure will be used to assess the exploratory hypothesis that the ESD violence prevention training will produce reductions in rates of exposure to gender-related violence. At baseline, participants will indicate whether they have been exposed to a list of gender-related victimization experiences since the age of 18. At the 3- and 6- month post-intervention followup, participants will indicate whether they have been exposed to these experiences "since your last assessment." Sample items include "I have been threatened with physical harm because of my gender identity or expression." "I have been pushed, shoved, hit, or had somethin thrown at me because of my gender identity or expression." Higher scores indicate greater exposure to gender-related violence. A likelihood of victimization score was calculated based on the average response to all measures on this subscale ("yes" vs "no"). Range: 0-1
Time Frame: Baseline
Population: A likelihood of victimization score was calculated based on the average response to all measures on this subscale ("yes" vs "no") among all participants who provided responses to at least two of the items on this scale. Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 35
score on a scale | .92 (1.54)

25. Secondary Outcome: Change in Endorsement of Gender-Based Victimization From Baseline to 3 Month Follow up
Description: as for outcome 24
Time Frame: Change from Baseline at 3 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 1 (1.45)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .38, t-test, 1 sided; Mean Difference (Net) = -.08, Standard Deviation 1.68

26. Secondary Outcome: Change in Endorsement of Gender-Based Victimization From Baseline to 6 Month Follow up
Description: as for outcome 24
Time Frame: Change from Baseline at 6 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
Number analyzed (Participants) | 36
score on a scale | 1.12 (1.85)
Statistical Analysis 1: Comparison: Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial; A one-tailed paired samples T-test was conducted to determine whether the post-treatment (i.e., 6-month) mean was statistically different from the baseline mean; Test type: Other; p = .25, t-test, 1 sided; Mean Difference (Net) = -.265, Standard Deviation 2.21

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants across each of the three groups received the same active treatment and were therefore assigned to a single treatment arm.
Arm/Group | Empowerment Self-Defense Training- Pre-Post Single Arm Design Pilot Trial
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT04934189/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04934189/SAP_003.pdf
  • Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT04934189/ICF_004.pdf